CLINICAL TRIAL: NCT05226572
Title: Repeated EUS-guided Fine Needle Biopsy of Pancreatic Masses After Non-diagnostic or Inconclusive Results - The REuBio Study
Brief Title: Repeated EUS-guided Fine Needle Biopsy of Pancreatic Masses After Non-diagnostic or Inconclusive Results
Acronym: REuBio
Status: Completed | Type: Observational
Sponsor: University of Bologna (Other)
Responsible Party: Principal Investigator, Pietro Fusaroli, Clinical Professor, University of Bologna
Other Study IDs: IMO-01
Record Dates: First submitted 2022-01-25; First posted 2022-02-07 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Pancreatic Adenocarcinoma; Pancreas Cancer; Pancreas Metastases
Keywords: Endoscopic Ultrasound; EUS-FNB; Solid Pancreatic lesion
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: endoscopic ultrasound-guided fine needle biopsy — repeated endoscopic ultrasound-guided fine needle-biopsy after a previous non diagnostic or incoclusive endoscopic ultrasound-guided tissue aquisition for pancreatic solid lesions.

SUMMARY:
The primary aim of REuBio study is to evaluate the diagnostic accuracy of repeated endoscopic ultrasound-guided fine needle biopsy after a previous non-diagnostic or inconclusive EUS-guided sampling of solid pancreatic lesions.

DETAILED DESCRIPTION:
Endoscopic ultrasound-guided fine needles biopsy (EUS-FNB) represents the gold standard method for the diagnosis of solid pancreatic lesions (SPLs), even if a non-negligible risk of false-negative or inconclusive results still exists.

In such cases, major guidelines recommend repeating EUS-guided tissue sampling. Nevertheless, this recommendation is not based on high-quality evidence and little is known about the performance of repeated EUS-FNB (rEUS-FNB).

The primary aim of this study is to evaluate the diagnostic accuracy of rEUS-FNB after a previous non-diagnostic or inconclusive EUS-guided sampling of SPLs.

The secondary aims of this study are to evaluate rEUS-FNB sensitivity, specificity, positive predictive value, negative predictive value, specimen adequacy, Bethesda classification, adverse events incidence and factors that influenced rEUS-FNB performance.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years old
* Solid pancreatic mass
* Previous non diagnostic or inconclusive EUS-tissue aquisition

Exclusion Criteria:

* age < 18 years old
* pancreatic mass with a predominantly cystic component
* previous pancreatic tissue acquisition was not performed under EUS-guidance (e.g. percutaneous sampling under abdominal ultrasound-guidance)
* repetition of pancreatic tissue sampling, after an inconclusive or non-diagnostic result, obtained by other methods than EUS-FNB, such as EUS-FNA or surgery or percutaneous sampling.
* patients with anatomic alterations or hematologic instability (including presence of severe blood clotting disorders) were excluded.
* rEUS-FNB of an extra-pancreatic mass

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A multicenter retrospective observational study enrolling all the consecutive patients who underwent a repeated EUS-guided tissue sampling for solid pancreatic masses with an EUS-FNB needle, after previous non-diagnostic or inconclusive result.
Sampling Method: Non-Probability Sample
Enrollment: 462 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2022-05-23 (Actual); Study Completion 2022-05-23 (Actual)

PRIMARY OUTCOMES:
Diagnostic yield (%) of repeated EUS-fine needle biopsy of pancreatic masses after previous non-diagnostic or inconclusive results | 5 years
  Outcome was measured as percentage (%)

SECONDARY OUTCOMES:
Sensitivity (%), specificity(%), positive predictive value(%), negative predictive value(%), specimen adequacy(%), Bethesda classification, adverse events incidence (%) and factors that influenced repeated EUS-fine needle biopsy performance. | 5 years
  Outcome was measured as percentage (%)

CONTACTS AND LOCATIONS:
Overall Officials: Pietro Fusaroli, Professor, Principal Investigator — University of Bologna
Locations (1):
- Gastrointestinal Unit, University of Bologna/Hospital of Imola, Bologna, Italy

IPD SHARING:
Plan to Share IPD: Undecided